CLINICAL TRIAL: NCT05386368
Title: Application of RECELL to Promote Healing Following CO2 Laser Treatment in Cosmetic Facelift Patients
Brief Title: RECELL to Promote Healing Following Carbon Dioxide (CO2) Laser Treatment in Cosmetic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. PI decided to terminate due to slow enrollment.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00085278
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Carbon Dioxide Laser; Photoaging
Keywords: Laser; Facelift

STUDY DESIGN:
Intervention Model Description: The perioral area of the face will be treated with CO2 laser. Laser setting will be determined by the treating surgeon for each individual patient - . The patient would be randomized and blinded to either left perioral or right perioral RECELL application - The surgeon would also be blinded to which side received RECELL treatment or Placebo (saline spray)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient would be randomized and blinded to either left perioral or right perioral RECELL application. The surgeon would also be blinded to which side received RECELL treatment or Placebo (saline spray).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Right receives ReCell (A) (Other): Right perioral area of face receives ReCell/ Left receives saline
  Interventions: Drug: ReCell
- Left receives ReCell (B) (Other): Left perioral area of face receives ReCell/ Right receives saline
  Interventions: Drug: ReCell

INTERVENTIONS:
Drug: ReCell — The perioral area of the face will be treated with CO2 laser. Randomization would occur before study initiation with subjects assigned either left perioral or right perioral RECELL treatment based on their subject enrollment number. The study team member who prepares and blinds the RECELL will create the list of subject ID numbers with subject ID number randomly assigned to either left perioral or right perioral treatment group. This will be completed prior to any patient enrollment in the study. Intraoperatively, RECELL and Placebo will be provided to surgeons and assistants in opaque application devices prepared by a trained, designated study team member.
  Both the treatment and placebo sides, will be dressed with a standard autologous cell suspension post treatment dressing (Telfa Clear and Xeroform).
  Other Names: autologous cell harvesting

SUMMARY:
To determine whether following Carbon dioxide (CO2) laser treatment, application of autologous cell suspension obtained via enzymatic and mechanical preparation will reduce negative side effects from CO2 laser and decrease the time of healing following treatment.

DETAILED DESCRIPTION:
The perioral area of the face will be treated with CO2 laser. Laser setting will be determined by the treating surgeon for each individual patient. Typical settings to be used for severe facial photoaging is Energy (mj) 100-125, Scan Size 6-7 mm, Density 2-3, Hertz 100-200, Repeat Delay 0.3-1.5 seconds, number of passes 2. The patient would be randomized and blinded to either left perioral or right perioral RECELL application. The surgeon would also be blinded to which side received RECELL treatment or Placebo (saline spray). Randomization would occur before study initiation with subjects assigned either left perioral or right perioral RECELL treatment based on their subject enrollment number. The study team member who prepares and blinds the RECELL will create the list of subject ID numbers with subject ID number randomly assigned to either left perioral or right perioral treatment group. This will be completed prior to any patient enrollment in the study. This spreadsheet will be password protected and only accessible to study coordinators and the team member responsible for preparing RECELL.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Patients undergoing facelift with perioral CO2 laser treatment
* Skin that is Fitzpatrick Score 1 or 2

Exclusion Criteria:

* Prior perioral CO2 laser resurfacing
* Allergy to components of preparation system

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Molnar, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing individual participant data with other researchers at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Receives ReCell (A): Right perioral area of face receives ReCell/ Left receives saline
  ReCell: The perioral area of the face will be treated with CO2 laser. Randomization would occur before study initiation with subjects assigned either left perioral or right perioral RECELL treatment based on their subject enrollment number. The study team member who prepares and blinds the RECELL will create the list of subject ID numbers with subject ID number randomly assigned to either left perioral or right perioral treatment group. This will be completed prior to any patient enrollment in the study. Intraoperatively, RECELL and Placebo will be provided to surgeons and assistants in opaque application devices prepared by a trained, designated study team member.
  Both the treatment and placebo sides, will be dressed with a standard autologous cell suspension post treatment dressing (Telfa Clear and Xeroform).
- Left Receives ReCell (B): Left perioral area of face receives ReCell/ Right receives saline
  ReCell: The perioral area of the face will be treated with CO2 laser. Randomization would occur before study initiation with subjects assigned either left perioral or right perioral RECELL treatment based on their subject enrollment number. The study team member who prepares and blinds the RECELL will create the list of subject ID numbers with subject ID number randomly assigned to either left perioral or right perioral treatment group. This will be completed prior to any patient enrollment in the study. Intraoperatively, RECELL and Placebo will be provided to surgeons and assistants in opaque application devices prepared by a trained, designated study team member.
  Both the treatment and placebo sides, will be dressed with a standard autologous cell suspension post treatment dressing (Telfa Clear and Xeroform).
Period: Overall Study
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We only had one subject total and she received (A) Right receives Recell
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 71 [71 to 71] |  | 71 [71 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Sensitivity Scores - Redness
Description: surveys will be given to address redness - a scale of "not at all, A little, moderately, or extremely" Scale is, "not at all", "a little", "moderately", "extremely"
Time Frame: month 3
Population: We did not have any subjects that received (B) Left receives Recell
Measure: Number; unit: # of participants reporting not at all
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
# of participants reporting not at all | 1 |

2. Primary Outcome: Change in Skin Sensitivity Scores - Sensitivity to Light
Description: surveys will be given to address sensitivity to light - a scale of "not at all, A little, moderately, or extremely" Score is, "not at all", "a little", "moderately", "extremely"
Time Frame: month 3
Population: We did not have any subjects that received (B) Left receives Recell
Measure: Number; unit: # of participants reporting not at all
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
# of participants reporting not at all | 1 |

3. Primary Outcome: Change in Skin Sensitivity Scores - Tightness
Description: surveys will be given to address tightness - a scale of "not at all, A little, moderately, or extremely"
Time Frame: month 3
Population: We did not have any participants receive (B) Left receives ReCell
Measure: Number; unit: # of participants reporting not at all
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
# of participants reporting not at all | 1 |

4. Primary Outcome: Change in Skin Sensitivity Scores - Itching
Description: surveys will be given to address itching - a scale of "not at all, A little, moderately, or extremely"
Time Frame: month 3
Population: We did not have any participants receive (B) Left receives ReCell
Measure: Number; unit: # of participants reporting not at all
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
# of participants reporting not at all | 1 |

5. Primary Outcome: Change in Skin Sensitivity Scores - Burning
Description: surveys will be given to address burning - a scale of "not at all, A little, moderately, or extremely"
Time Frame: month 3
Population: We did not have any participants receive (B) left receives ReCell
Measure: Number; unit: # of participants reporting not at all
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
# of participants reporting not at all | 1 |

6. Primary Outcome: Change in Wong-Baker FACES Pain Assessment Tool Scores
Description: Wong-Baker FACES Pain Rating Scale - 1-10 pain scale - the higher the score the more pain
Time Frame: Month 3
Population: We did not have any participants receive (B) Left receives ReCell
Measure: Number; unit: score on a scale
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
score on a scale | 0 |

7. Secondary Outcome: Healing Within 2 Weeks Post-op
Description: Quantificare LifeViz Camera will be used - yes/no whether healing occurred within first 2 weeks post-op
Time Frame: month 3
Population: We did not have any participants receive (B) left receives ReCell
Measure: Number; unit: percentage of participants with healing
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
Number analyzed (Participants) | 1 | 0
percentage of participants with healing | 100 |

ADVERSE EVENTS:
Time Frame: 3 months
Description: We did not have any participants randomized to receive ReCell on the Left side, so there were no participants at risk in this arm.
Arm/Group | Right Receives ReCell (A) | Left Receives ReCell (B)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT05386368/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT05386368/ICF_002.pdf